CLINICAL TRIAL: NCT02545946
Title: Traditional Incision and Drainage of Cutaneous Abscess Vs. Minimally Invasive Incision and Drainage With Vessel Loop: A Randomized Control Trial.
Brief Title: Trial of Abscess Drainage Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00033369
Record Dates: First submitted 2015-07-29; First posted 2015-09-10 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Cutaneous Abscess
Keywords: traditional incision and drainage; minimally invasive incision and drainage; vessel loop; emergency department; pediatrics
MeSH Terms: conditions — Emergencies | interventions — Drug Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional (Active Comparator): cutaneous abscess with be opened in the traditional incision and drainage technique with large incision, breaking up of pockets of pus, washing out the pocket and with or without packing gauze placed into residual cavity
  Interventions: Other: traditional I&D with or without packing
- Minimally Invasive (Active Comparator): Cutaneous abscess will be opened with two small incisions just large enough to pass a vessel loop through both to keep them open. Pockets of pus will be broken up and the cavity washed out before placing the loop through both incisions and loosely tieing it over the skin
  Interventions: Device: vessel loop

INTERVENTIONS:
Device: vessel loop — using the vessel loop to hold the place of the surgical wound that is made during I&D
  Arms: Minimally Invasive
Other: traditional I&D with or without packing — abscess will be drained with a traditional I&D with or without packing (as deemed appropriate by ER doctor)
  Arms: Traditional

SUMMARY:
Comparing the outcome of traditional incision and drainage with a larger skin incision with or without gauze packing of cutaneous abscess in pediatrics versus a new minimally invasive incision and drainage with two small incisions and a vessel loop transversing the incisions to keep them open.

DETAILED DESCRIPTION:
This prospective randomized single blind clinical trial will be conducted in a suburban pediatric emergency department that treats approximately 29,000 patients per year. Patients between 0-17 years with a superficial skin or soft tissue abscess larger than 3 cm that would be appropriate for ED I&D and outpatient management will be screened for inclusion. Patients will be excluded if they are immunocompromised (taking chemotherapy, steroid or bioactive medications or having diabetes mellitus), require a subspecialist for drainage or require hospitalization. Subjects will be required to provide assent when age-appropriate, and parental consent will be obtained. The parent or guardian will need to be in the emergency department with the child to provide consent. Subjects will be randomized to be in either the traditional I&D arm or the minimally invasive vessel loop arm using numbered sealed envelops. Computer blocking will randomize these numbered envelopes. Inside the envelope there will be instructions to the treating physician as to which of two standard techniques should be employed.

* Standardized I&D will be performed with a #11 blade scalpel and a full thickness cut incising the lesion along at least 50% of the abscess diameter. The pocket will then be probed to break up septations and the residual cavity will be irrigated with normal saline. Iodinated gauze 0.25 inch will be used to loosely pack the remaining cavity if the physician deems packing is necessary. The gauze will be left trailing out of the surgical incision. The abscess will then be covered with 4 X 4 dry gauze and taped in place.
* Minimally invasive I&D with vessel loop will be preformed by making a 5mm incision with a #11 blade in the area of maximal fluctuance. The cavity will then be probed with forceps breaking up any septations. The forceps will then be used to find the furthest extent of the cavity, and the #11 blade will be used to make a 5mm incision at the tip of the forceps (at the farthest extent of the cavity). The forceps will then be pushed through this second incision. The vessel loop will be grasped by the forceps and then pulled back through both surgical incisions. The vessel loop will then be tied loosely together, creating a loop back through both surgical incisions. Both sides of the incisions will then be irrigated with normal saline.

Cultures will be obtained, if possible, from the abscess. Pain medication and sedation at the time of the I&D will be left to the discretion of the treating physician. Antibiotics will not be mandated, but allowed at the judgment of the treating medical team. All subjects will be given 2 prescriptions for analgesia at home. One for mild pain, ibuprofen; another for moderate or severe pain, acetaminophen with hydrocodone (either liquid or pills) will be given. Equipotent alternatives will be provided in case of medication allergy. Pain scores will be assessed using a ten point scale before and after the procedure and at 48 hour follow up. Data recorded at the first visit will include demographics (age, male/female), characteristics of the abscess, fever, duration of symptoms, history of prior abscess, antibiotics in the last month, and provision of antibiotics post-procedure.

All subjects will return to the ER in 72 hours and 1 week for a recheck. At the 3rd day visit, wound packing will be removed. Large cavities will be repacked at the discretion of the ED physician. Loops will be cut and removed at the 7th day visit unless significant cellulitis remains. If cellulitis remains after 7 days, additional visits/hospitalization would be set up at the treating doctors discretion. Given that failure of treatment is a possible event in any abscess drainage, even those not involved with this study, hospitalization or additional visits beyond the 2 included in the study, will be billed to the patient's family and/or insurance company as any visit to the ER or hospital admission.

Patients and families will also be contacted at one month via telephone interview. Self-rated cosmetic outcome will be assessed using a 10 point scale from worst to best looking scar.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient (0-18 years old) with abscess over 3 cm which can be drained in the ER and does not require hospitalization

Exclusion Criteria:

* Diabetes
* immunocompromised
* cancer
* chemotherapy
* requires hospitalization for treatment of abscess
* abscess felt not drainable in the ER by ER physicians

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-07-07 (Actual)

PRIMARY OUTCOMES:
number of patients who require repeat I&D collected by data form | 1 week
  any patient that needs an additional I&D procedure noted on data collection forms
Number of patients who Need to have an antibiotic added to treatment plan/or changed antibiotic after the initial visit collected by data form | 1 week
  any patient requiring the above noted on data collection forms
the number of patients who need to be hospitalized after the first visit collected by data form | 1 week
  if patient is hospitalized after first visit, as collected on data form

SECONDARY OUTCOMES:
patient satisfaction with procedure collected by survey | 1 day
  1-100 scale of satisfaction survey with the drainage performed
patient satisfaction with healing of abscess collected by survey | 1 month
  1-100 scale survey of how satisfied patient is with how the drainage site healed
patient satisfaction with overall treatment of the abscess collected by survey | 1 month
  1-100 scale survey for how satisfied patient is with overall care related to abscess

CONTACTS AND LOCATIONS:
Overall Officials: Milan Nadkarni, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided